CLINICAL TRIAL: NCT03417726
Title: "Evaluation of Pediatric Balance Scale and Quantitative Balance Parameters in Patients With Cerebral Palsy"
Brief Title: Evaluation of Pediatric Balance Scale and Quantitative Balance Parameters in Patients With Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2017.735
Record Dates: First submitted 2018-01-11; First posted 2018-01-31 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Cerebral Palsy, Spastic; Balance; Distorted
Keywords: Cerebral Palsy; Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate Pediatric Balance Scale and quantitative balance and gait parameters assessed by Balance Master force plate in Cerebral Palsy (CP) patients who are ambulatory without an assistive device in daily life.

DETAILED DESCRIPTION:
CP refers to a group of motion and posture disorders that limit activity and participation which is attributed to non-progressive disturbances in the developing fetus or infant brain. In CP, motor and sensory disorders are often accompanied by poor balance control. Impaired balance control leads to increased risk of falling, which is a major kinesiologic problem in children who are ambulatory without an assistive device.

Functional balance in children is defined as the ability to maintain the center of gravity according to the base of support during typical childhood activities of daily living, school and play. The Pediatric Balance Scale, a modification of the Berg Balance Scale, was developed as a functional balance measure for children, easily administered without specialized equipment in a relatively short time.

Balance Master® (Neurocom International Clackmas, Oregon, USA) is a device consisting of a system that processes signals from an 18x60 inch plaque that transmits the vertical forces exerted through patient's feet to measure center of gravity position and postural control through a software program.

The aim of this study is to compare PBS results with quantitative balance and gait parameters obtained from Balance Master in spastic CP patients who are independently ambulatory. The level of correlation between these measurement methods will be examined and superiority to each other in assessing balance problems in this patient group will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with spastic cerebral palsy
* Age between 4-18 years
* Sufficient cooperation to understand instructions and participate evaluations
* Gross Motor Function Classification System (GMFCS) level I-II
* Giving an informed consent

Exclusion Criteria:

* Visual and vestibular deficits
* Botulinum-toxin A treatment within 3 months or having undergone an orthopaedic surgery 1 year prior to inclusion in the study
* Severe scoliosis (Cobb angle >40°)
* Uncontrolled seizures (Seizure in previous 6 months)
* Having intrathecal baclofen pump
* Having undergone selective dorsal rhizotomy

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Spastic Cerebral Palsy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) - Firm-Eyes Open | 2 min
  Evaluations will be done by Balance Master® (Neurocom International Clackmas, Oregon, USA) device which consists a system that processes signals from an 18x60 inch plaque that transmits the vertical forces exerted through patient's feet to measure center of gravity (COG) position and postural control through a software program. Each assessment will be made 3 times and average scores will be calculated via program.
  Mean COG Sway Velocity (deg/sec) during standing on a Firm Surface-Eyes Open is the primary outcome measure.

SECONDARY OUTCOMES:
Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) - Firm-Eyes Closed, Foam-Eyes Open, Foam-Eyes Closed | 3 min
  Evaluations will be done by Balance Master® (Neurocom International Clackmas, Oregon, USA) device which consists a system that processes signals from an 18x60 inch plaque that transmits the vertical forces exerted through patient's feet to measure center of gravity position and postural control through a software program. Each assessment will be made 3 times and average scores will be calculated via program.
  Mean COG Sway Velocity (deg/sec) and COG Alignment during 3 sensory conditions will be assessed as secondary outcome measures: Firm-Eyes Closed, Foam-Eyes Open, Foam-Eyes Closed.
Limits of Stability (LOS) | 2 min
  Evaluations will be done by Balance Master® device. Reaction Time (sec), Movement Velocity (deg/sec), Endpoint Excursions (%), Max Excursions (%) and Directional Control (%) will be recorded during forward leaning.
Walk Across (WA) | 5 min
  Evaluations will be done by Balance Master® device. Gait parameters; Step Width (cm), Step Length (cm), Speed (cm/sec), Step Length Symmetry (%) will be recorded while walking across the forceplate. Each assessment will be made 3 times and average scores will be calculated via program.
Tandem Walk (TW) | 5 min
  Evaluations will be done by Balance Master® device. Step Width (cm), Speed (cm/sec), End Sway (deg/sec) will be recorded as the patient walks heel to toe from one end of the forceplate to the other as quickly as possible and then stop. Each assessment will be made 3 times and average scores will be calculated via program.
Unilateral Stance (US) | 5 min
  Evaluations will be done by Balance Master® device. Mean COG Sway Velocity (deg/sec) will be recorded during left and right single leg standing while eyes open. Each assessment will be made 3 times and average scores will be calculated via program.
Step/Quick Turn (SQT) | 5 min
  Evaluations will be done by Balance Master® device. Turn Time (sec), Turn Sway (deg), Left/Right Turn Time Difference (%) and Left/Right Turn Sway Difference (%) will be recorded as the patient walks from one end of the forceplate to the other, take a quick 180 degrees turn to either left or right and return to the starting point. Each assessment will be made 3 times and average scores will be calculated via program.
Pediatric Balance Scale (PBS) | 20 min
  PBS is a functional balance scale adapted and customized from Berg Balance Scale for use with children. The PBS has been used initially to measure the balance functions for school-age children with mild-to-moderate motor impairments. A recent study has shown that PBS is also sensitive in assessing functional balance differences in children aged 4-10 with a rough motor function classification system (KMFSS) level 1-2
  The PBS is a 14-item, criterion-referenced measure, which examines functional balance in the context of everyday tasks. It can easily be administered and scored in less than 20 minutes using equipment commonly found in schools and clinics. Scoring (0-4) is based on how long a specific movement or position is performed, how long the position can be maintained, or how much assistance it requires. The highest score in PBS is 56.
Selective Control Assessment of the Lower Extremity (SCALE) | 15 min
  The SCALE tool was designed for clinical administration and scoring by healthcare professionals, to be used in less than 15 minutes without specialized equipment. The tool includes 'Directions for Administration,' 'Instructions for Grading,' and a 'Score Sheet.' Hip, knee, ankle, subtalar, and toe joints are assessed bilaterally. The following factors were used to develop the assessment and grading criteria: (1) ability to move each joint selectively; (2) involuntary movement at other joints including the contralateral limb; (3) ability to reciprocate movement; (4) speed of movement; and (5) generation of force as demonstrated by excursion within the available range of motion. Selective voluntary motor control is graded at each joint as 'Normal' (2 points), 'Impaired' (1 point), or 'Unable' (0 points).

CONTACTS AND LOCATIONS:
Overall Officials: Naime Evrim Karadag Saygi, Prof, Study Chair — Marmara University School of Medicine, Pendik Research and Training Hospital, Department of Physical Medicine and Rehabilitation, Istanbul / Turkey 34890
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Fowler EG, Staudt LA, Greenberg MB, Oppenheim WL. Selective Control Assessment of the Lower Extremity (SCALE): development, validation, and interrater reliability of a clinical tool for patients with cerebral palsy. Dev Med Child Neurol. 2009 Aug;51(8):607-14. doi: 10.1111/j.1469-8749.2008.03186.x. Epub 2009 Feb 12. PMID 19220390
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Saether R, Helbostad JL, Riphagen II, Vik T. Clinical tools to assess balance in children and adults with cerebral palsy: a systematic review. Dev Med Child Neurol. 2013 Nov;55(11):988-99. doi: 10.1111/dmcn.12162. Epub 2013 May 16. PMID 23679987